CLINICAL TRIAL: NCT04843501
Title: Middle School Cluster RCT to Evaluate E-Cigarette Prevention Program: CATCH My Breath
Brief Title: Middle School Cluster Randomized Controlled Trial (RCT) to Evaluate E-Cigarette Prevention Program: CATCH My Breath
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Steven H. Kelder, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC-SPH-18-0254; 5R01CA242171-02 (NIH)
Record Dates: First submitted 2021-04-08; First posted 2021-04-13 (Actual); Results first posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: E-cigarette Use
Keywords: E-cigarette Prevention
MeSH Terms: conditions — Vaping | interventions — Tea

STUDY DESIGN:
Intervention Model Description: 10 schools will receive the experimental CATCH My Breath program and 10 schools will receive the usual care Texas Education Agency required tobacco prevention program. Each school will include 70 students.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CATCH My Breath (CMB) program for E-cigarette prevention among adolescents (Experimental): The CMB curriculum is divided into four developmentally appropriate e-cigarette lessons (approximately 20-30 minutes each) for middle school aged youth (6th - 8th grade). A variety of educational strategies are used and include cooperative learning groups, large group discussions, interviews, role-play, media, reports, and goal setting. CMB will provide study materials to teachers and schools through a state-of-the art online delivery portal. A site-based management team will oversee program implementation. Teachers will be trained via webinar. Project staff will visit all participating schools to assemble and train the CATCH site-based management team, and answer questions about the study. Teachers in CMB intervention schools will be provided with CMB-specific training for implementing the lessons with fidelity through a one-hour live webinar with Dr. Kelder, which will be offered at multiple times to accommodate teaching schedules.
  Interventions: Behavioral: CATCH My Breath (CMB) program for E-cigarette prevention among adolescents
- Texas Education Agency required tobacco prevention program (Active Comparator): The TEA tobacco prevention program is a state-supported program that meets the mandates of the state. It includes online lessons and support materials.
  Interventions: Behavioral: Texas Education Agency (TEA) required tobacco prevention program

INTERVENTIONS:
Behavioral: CATCH My Breath (CMB) program for E-cigarette prevention among adolescents — CMB has 4 developmentally appropriate e-cigarette lessons, 20-30 minutes in each of 6th-8th grades. Strategies include small and large group discussions, parent interviews, role-plays, media literacy, and goal setting. E-cigarette focused science and humanities activities (2 per school year) are also provided. An informational tool kit will be provided to parents. Finally, 8 activity-based E-cig PE lessons are intended for either 7th or 8th grades, depending on school calendar. CMB provides study materials to teachers through an online access portal. A site-based management team will oversee program implementation. Teachers in CMB intervention schools will be provided with CMB-specific training for implementing the lessons with fidelity through a one-hour live webinar, offered at multiple times to accommodate teaching schedules. Project staff will meet routinely with participating schools to answer study questions.
  Arms: CATCH My Breath (CMB) program for E-cigarette prevention among adolescents
Behavioral: Texas Education Agency (TEA) required tobacco prevention program — The TEA tobacco prevention program is a state-supported program that meets the mandates of the state. It includes TEA developed online lessons and support materials and also includes elements of the CDC Know the Risks e-cigarette prevention program. This can be considered 'usual care'
  Arms: Texas Education Agency required tobacco prevention program

SUMMARY:
This is a two-arm, cluster randomized trial designed to to evaluate the effectiveness of an e-cigarette curriculum [called the CATCH My Breath (CMB) program] in delaying the onset of e-cigarette use in middle schoolers. Schools will be assigned to either the CMB program or usual care, which is Texas Education Agency (TEA) required tobacco prevention program. 10 schools will be assigned to each arm arm, and each school will include 70 students in the study, for a total of 700 students per arm and 1400 total students in the study. Both programs will be administered to participating students over 3 years.

DETAILED DESCRIPTION:
The goal of this research is to empirically assess the three year immediate effects and 12 year follow-up of the CATCH My Breath (CMB) program on delaying the onset of e-cigarette use with a 6th-9th grade cohort, using a 20-school group randomized controlled trial (RCT), with 1,400 students. E-cigarettes are the most commonly used tobacco product by US youth. Recent research, strongly suggests that youth who only smoke e-cigarettes exhibit symptoms of addiction, and are more likely to experiment combustible tobacco. Unfortunately, few e-cigarette prevention programs exist, and none have been tested for longer-term efficacy. Although some tobacco prevention programs have included an e-cigarette add -on component, to our knowledge, none of these revised programs have been formally evaluated. The lack of e-cigarette specific program content, and lack of rigorous evaluation, warrants the proposed project. CMB was developed with input from school administrators, health education coordinators, tobacco prevention educators, classroom teachers, students, and parents. CMB has been formatively evaluated and pilot tested at 59 middle schools in 7 states, resulting in positive feedback from over 100 middle school teachers and 9,578 6th-8th grade students. Our second pilot pretest-posttest controlled experiment (2017-2018), and resulted in an treatment-control difference of 3.8% in ever smoking over a 16-month period. Given CMB's current popularity with schools as a 'best practice' program, and with initial positive results, a full scale randomized control trial is needed to determine longer term, 6th-9th grade efficacy.

ELIGIBILITY:
School Inclusion Criteria:

* enrollment of at least 70 students in each of the 6th, 7th, and 8th grades
* school location is 100 miles of research site

School Exclusion Criteria:

* schools that have participated in the previous 2 pilot tests
* currently implementing CMB

Student Inclusion Criteria:

* enrollment in the 6th grade at a study school
* willingness to complete the measurements six times during the study

Student Exclusion Criteria:

- severe disabilities that limit their participation

Parent Inclusion Criteria:

* ability to communicate in English or Spanish
* caretaker of a 6th-grade child.

Parent Exclusion Criteria:

-inability to communicate in English or Spanish

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2059 (Actual)
Dates: Start 2020-12-13 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven H Kelder, PhD, MPH, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston School of Public Health at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 2059 participants enrolled in the study, 5 participants withdrew before starting the study. Eligible individuals could enroll at the start of any semester. Participation was not required to be continuous, and participant numbers varied by semester.
Units Other Than Participants: Schools
Groups:
- CATCH My Breath (CMB) Program for E-cigarette Prevention Among Adolescents: CATCH My Breath (CMB) program for E-cigarette prevention among adolescents: CMB has 4 developmentally appropriate e-cigarette lessons, 20-30 minutes in each of 6th-8th grades. A variety of educational strategies are used and include cooperative learning groups, large group discussions, interviews, role-play, media, reports, and goal setting. E-cigarette focused science and humanities activities (2 per school year) are also provided. An informational tool kit will be provided to parents. Finally, 8 activity-based E-cig PE lessons are intended for either 7th or 8th grades, depending on school calendar. CMB will provide study materials to teachers and schools through a state-of-the art online delivery portal. A site-based management team will oversee program implementation. Teachers will be trained via webinar. Project staff will visit all participating schools to assemble and train the CATCH site-based management team, and answer questions about the study. Teachers in CMB intervention schools will be provided with CMB-specific training for implementing the lessons with fidelity through a one-hour live webinar with Dr. Kelder, which will be offered at multiple times to accommodate teaching schedules.
Period: Fall 2021
Arm/Group | CATCH My Breath (CMB) Program for E-cigarette Prevention Among Adolescents | Texas Education Agency Required Tobacco Prevention Program
Started | 1110; 12 Schools | 611; 10 Schools
Completed | 1110; 12 Schools | 611; 10 Schools
Not Completed | 0; 0 Schools | 0; 0 Schools
Period: Spring 2022
Arm/Group | CATCH My Breath (CMB) Program for E-cigarette Prevention Among Adolescents | Texas Education Agency Required Tobacco Prevention Program
Started (Of the 1110 students who enrolled in Fall 2021 in the CATCH My Breath (CMB) program for E-cigarette prevention among adolescents arm, 180 students were added and 398 students left resulting in 892 students enrolled in Spring 2022. Of the 611 students who enrolled in Fall 2021 in the Texas Education Agency required tobacco prevention program arm, 59 students were added and 213 students left resulting in 457 students enrolled in Spring 2022.) | 892; 12 Schools | 457; 10 Schools
Completed | 892; 12 Schools | 457; 10 Schools
Not Completed | 0; 0 Schools | 0; 0 Schools
Period: Fall 2022
Arm/Group | CATCH My Breath (CMB) Program for E-cigarette Prevention Among Adolescents | Texas Education Agency Required Tobacco Prevention Program
Started (Of the 892 students who started in Spring 2022 in the CATCH My Breath (CMB) program for E-cigarette prevention among adolescents arm, 26 students were added and 59 students left resulting in 859 students enrolled in Fall 2022. Of the 457 students who started in Spring 2022 in the Texas Education Agency required tobacco prevention program arm, 18 students were added and 69 students left resulting in 406 students enrolled in Fall 2022.) | 859; 12 Schools | 406; 10 Schools
Completed | 859; 12 Schools | 406; 10 Schools
Not Completed | 0; 0 Schools | 0; 0 Schools
Period: Spring 2023
Arm/Group | CATCH My Breath (CMB) Program for E-cigarette Prevention Among Adolescents | Texas Education Agency Required Tobacco Prevention Program
Started | 898; 12 Schools | 434; 10 Schools
Completed | 898; 12 Schools | 434; 10 Schools
Not Completed | 0; 0 Schools | 0; 0 Schools
Period: Fall 2023
Arm/Group | CATCH My Breath (CMB) Program for E-cigarette Prevention Among Adolescents | Texas Education Agency Required Tobacco Prevention Program
Started | 755; 12 Schools | 412; 10 Schools
Completed | 755; 12 Schools | 412; 10 Schools
Not Completed | 0; 0 Schools | 0; 0 Schools
Period: Spring 2024
Arm/Group | CATCH My Breath (CMB) Program for E-cigarette Prevention Among Adolescents | Texas Education Agency Required Tobacco Prevention Program
Started | 533; 12 Schools | 301; 10 Schools
Completed | 533; 12 Schools | 301; 10 Schools
Not Completed | 0; 0 Schools | 0; 0 Schools

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CATCH My Breath (CMB) Program for E-cigarette Prevention Among Adolescents | Texas Education Agency Required Tobacco Prevention Program | Total
Number analyzed (Participants) | 1332 | 727 | 2059
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1332 | 727 | 2059
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 643 | 352 | 995
  Male | 672 | 364 | 1036
  Unknown or Not Reported | 17 | 11 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 784 | 388 | 1172
  Not Hispanic or Latino | 531 | 328 | 859
  Unknown or Not Reported | 17 | 11 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 22 | 14 | 36
  Asian | 52 | 31 | 83
  Native Hawaiian or Other Pacific Islander | 8 | 4 | 12
  Black or African American | 142 | 91 | 233
  White | 434 | 259 | 693
  More than one race | 175 | 105 | 280
  Unknown or Not Reported | 499 | 223 | 722
Region of Enrollment [Number; unit: participants]
  United States | 1332 | 727 | 2059

OUTCOME MEASURES:

1. Primary Outcome: Number of Students Who Currently Use E-cigarettes
Description: Current use is defined as e-cigarette use in the last 30 days.
Time Frame: baseline
Population: Participants who reported ever using e-cigarettes at baseline were included in the analysis for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | CATCH My Breath (CMB) Program for E-cigarette Prevention Among Adolescents | Texas Education Agency Required Tobacco Prevention Program
Number analyzed (Participants) | 37 | 17
Participants | 9 | 4

2. Primary Outcome: Number of Students Who Currently Use E-cigarettes
Description: Current use is defined as e-cigarette use in the last 30 days.
Time Frame: 3 years
Population: Participants who reported ever using e-cigarettes at 3 years were included in the analysis for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | CATCH My Breath (CMB) Program for E-cigarette Prevention Among Adolescents | Texas Education Agency Required Tobacco Prevention Program
Number analyzed (Participants) | 27 | 25
Participants | 5 | 1

3. Primary Outcome: Number of Students Who Have Ever Used E-cigarettes in Their Lifetime
Time Frame: baseline
Measure: Count of Participants; unit: Participants
Arm/Group | CATCH My Breath (CMB) Program for E-cigarette Prevention Among Adolescents | Texas Education Agency Required Tobacco Prevention Program
Number analyzed (Participants) | 1332 | 727
Participants | 37 | 17

4. Primary Outcome: Number of Students Who Have Ever Used E-cigarettes in Their Lifetime
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | CATCH My Breath (CMB) Program for E-cigarette Prevention Among Adolescents | Texas Education Agency Required Tobacco Prevention Program
Number analyzed (Participants) | 533 | 301
Participants | 27 | 25

5. Primary Outcome: Number of Students Who Are Susceptible to E-cigarette Use
Description: Susceptibility to e-cigarette use is defined as never used an e-cigarette but having tendencies that indicate that e-cigarette use is likely. Susceptibility is assessed with a questionnaire that asks "Do any of your friends use e-cigarettes?," "Are you curious about e-cigarettes?," and "Do you think you will try an e-cigarette in the next year?" Yes to any of these three questions indicates susceptibility to e-cigarette use.
Time Frame: baseline
Population: Participants who indicated they have never used an e-cigarette were assessed for this outcome. Data were only collected for participants who answered the questions.
Measure: Count of Participants; unit: Participants
Arm/Group | CATCH My Breath (CMB) Program for E-cigarette Prevention Among Adolescents | Texas Education Agency Required Tobacco Prevention Program
Number analyzed (Participants) | 1034 | 528
Participants | 357 | 171

6. Primary Outcome: Number of Students Who Are Susceptible to E-cigarette Use
Description: as for outcome 5
Time Frame: 3 years
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | CATCH My Breath (CMB) Program for E-cigarette Prevention Among Adolescents | Texas Education Agency Required Tobacco Prevention Program
Number analyzed (Participants) | 490 | 262
Participants | 171 | 95

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | CATCH My Breath (CMB) Program for E-cigarette Prevention Among Adolescents | Texas Education Agency Required Tobacco Prevention Program
All-Cause Mortality (participants affected / at risk) | 0/1332 | 0/727
Serious Adverse Events (participants affected / at risk) | 0/1332 | 0/727
Other Adverse Events (participants affected / at risk) | 0/1332 | 0/727

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/01/NCT04843501/Prot_SAP_000.pdf
  • Informed Consent Form (2018-06-20): https://cdn.clinicaltrials.gov/large-docs/01/NCT04843501/ICF_001.pdf